CLINICAL TRIAL: NCT03958201
Title: Best Management of Muscle Relaxation With Rocuronium Using Objective Monitoring and Reversal With Neostigmine or Sugammadex
Brief Title: Best Management of Muscle Relaxation- Objective Monitoring
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Washington (Other)
Responsible Party: Principal Investigator, Stephan Thilen, Assistant Professor, School of Medicine: Anesthesiology & Pain Medicine, University of Washington
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: STUDY00007084
Record Dates: First submitted 2019-05-17; First posted 2019-05-21 (Actual); Results first posted 2022-11-02 (Actual); Last update posted 2022-11-02 (Actual); Status verified 2022-10

CONDITIONS: Residual Paralysis, Post Anesthesia
MeSH Terms: conditions — Delayed Emergence from Anesthesia | interventions — Clinical Protocols; Neostigmine; Sugammadex

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Protocol (Other): Patients will have perioperative neuromuscular block managed by protocol. The protocol includes specified appropriate rocuronium dosing and reversal with either neostigmine or sugammadex depending on depth of block as assessed objectively at adductor pollicis with quantitative neuromuscular monitoring.
  Interventions: Combination Product: Protocol for Management of Muscle Relaxation With Rocuronium Using Objective Monitoring and Reversal With Neostigmine or Sugammadex

INTERVENTIONS:
Combination Product: Protocol for Management of Muscle Relaxation With Rocuronium Using Objective Monitoring and Reversal With Neostigmine or Sugammadex — The protocol includes specified appropriate rocuronium dosing and a valid pre-reversal assessment of the adductor pollicis response guides optimal neostigmine vs. sugammadex reversal.

SUMMARY:
The purpose of this study is to demonstrate that the investigators can reduce residual paralysis to a very low incidence, and that the investigators can do this while preserving a role for the older and less expensive reversal agent neostigmine. The investigators consider this an evidence-based approach because previous reports clearly indicate that neostigmine is effective for reversal of the most shallow neuromuscular blocks, a level of block now referred to as minimal block. The Investigators also know from previous data that a substantial proportion of patients have minimal block. Sugammadex will be used when the block to be reversed is deeper than minimal, specifically when the objectively measured TOF-ratio is <40%.

The investigators hypothesize that this protocol will be associated with an incidence of residual paralysis of less than 3%. The investigators plan is to study 200 patients.

DETAILED DESCRIPTION:
This study implements a standardized protocol for NMBD (neuromuscular blocking drug) management that is currently used by some providers at UWMC and HMC to help prevent residual paralysis in surgical patients. While this protocol is within the scope of routine care that an anesthesiologist could follow in his/her clinical practice, it is not consistently used throughout HMC and UWMC. This protocol follows clinical best practices for NMBD management in a surgical population and adheres to the recommendations from the P&T committee on reversal drug choice and recommendations from the Department of Anesthesiology and Pain Medicine on neostigmine dosing. While this protocol is in line with best practices, the investigators are continuing to systematically evaluate it in the setting of prospective research. All drugs will be administered for clinical care only. This research does not add additional medications. The study will take place at UWMC and HMC and will follow a standardized research protocol for the timing, dosing, and monitoring surrounding muscle relaxants and reversal, and makes use of objective TOF monitors. If a patient agrees to participate in this study, the following research protocol will occur:

Before Surgery:

1. TOF measurements before surgery: A study investigator will perform the routine clinical train-of-four measurements with an objective monitor at baseline after the clinical induction of general anesthesia but before the administration of the NMBD. Information will be recorded for research purposes. Research staff will leave the operating room after obtaining the baseline measurement and will return to the operating room at the end of the surgical procedure, to be available for TOF ratio measurements at the time that reversal of paralysis is planned as well as for the primary outcome measurement, i.e. at time of extubation.
2. Dose calculation of initial NMBD: A study investigator will assist the anesthesia provider with calculation of the recommended intubating dose of rocuronium (an NMBD). The dose will be calculated per this research protocol based on Ideal Body Weight (IBW).

   1. For women 45.5 kg plus 2.3 kg/inch over 5 feet of height
   2. For men 50 kg plus 2.3 kg/inch over 5 feet of height.
   3. For routine intubations, the recommended dose for intubation will be a maximum of Rocuronium 0.6 mg/kg.
   4. The intubating dose will be reduced by 15% for females.
   5. Higher intubating dose may be used at the discretion of the anesthesia provider

During Surgery:

1. Additional dose calculation of NMBD: Each additional dose of rocuronium will be 25% of the recommended intubating dose and will be administered when the TOF count has returned to at least 2, the aim is to maintain an intraoperative TOF count of 1-2 unless the anesthesia provider has deemed deep paralysis to be necessary in which case a TOF count of 0 will be maintained. An attempt will be made to avoid administration of rocuronium during the last 30 minutes of the procedure.

After Surgery:

1. Patients will receive reversal drugs for their routine care that will help reverse the effects of their muscle relaxant. In this study, the decision of reversal drug use will follow institutional guidelines. The timing and dose calculation of the reversal drug will follow the research protocol as follows:
2. Timing of neostigmine or sugammadex: Based on the results of the clinical pre-reversal TOF assessment, reversal with neostigmine will be administered if the objective TOF-ratio is between 40%-90%. If the block is deeper than this, then sugammadex will be used for reversal (This is per institutional guidance on choice of reversal drug).
3. Dose calculation of neostigmine and sugammadex: For this study, the dose of neostigmine will be calculated based on the IBW. The dose of sugammadex will be calculated based on patients' actual body weight.

   For all subjects enrolled in this study, the investigators will follow a dose schedule which is based on clinical TOF monitoring and is in accordance with institutional recommendations for dosing of neostigmine.
4. Timing of extubation: The patient's trachea will not be extubated before routine objective monitoring confirms recovery to a TOF-ratio 90%. However, in the case that objective monitoring cannot be obtained by the provider then the following will happen:

   1. For subjects who receive neostigmine for their routine care, it is recommended that the patient's trachea will not be extubated earlier than 10 minutes after the administration of this drug.
   2. For subjects who receive sugammadex for routine care, it is recommended that the patient's trachea will not be extubated earlier than 3 minutes after drug administration.
5. TOF measurements after surgery (extubation): The TOF-ratio will be measured by a study investigator or provider at the time of extubation. Information will be recorded for research purposes. If the investigators miss obtaining research measurements at the time of extubation, they will obtain TOF measurements on the patient's arrival to the PACU.
6. Collection of data from EMR: the investigators will collect information from the patient's medical record including the intraoperative TOF counts, ASA class, surgical procedure, times of the surgical procedure, time and dose of administered medications, and the patient's temperature in the operating room and PACU.

ELIGIBILITY:
Inclusion Criteria:

* Are 18 years or older
* Undergoing surgery expected to last less than 6 hours at HMC or UWMC
* Have ASA physical status I-III
* Scheduled to have general anesthesia with at least 1 dose of nondepolarizing NMBD for endotracheal intubation or intraoperative neuromuscular block (NMB)

Exclusion Criteria:

* Allergy to NMBDs, neostigmine, or sugammadex
* Patients with neuromuscular disease (myasthenia gravis or muscular dystrophy)
* Pregnant or lactating women
* Non English speaking
* Unable to provide informed consent
* Severe renal failure with eGFR less than 20 ml/min

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2019-05-28 (Actual); Primary Completion 2020-01-31 (Actual); Study Completion 2020-03-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stephan R Thilen, MD, Principal Investigator — University of Washington
Locations (1):
- Harborview Medical Center, Seattle, Washington, United States

REFERENCES:
- [Derived] Thilen SR, Sherpa JR, James AM, Cain KC, Treggiari MM, Bhananker SM. Management of Muscle Relaxation With Rocuronium and Reversal With Neostigmine or Sugammadex Guided by Quantitative Neuromuscular Monitoring. Anesth Analg. 2024 Sep 1;139(3):536-544. doi: 10.1213/ANE.0000000000006511. Epub 2023 May 12. PMID 37171989

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 200 subjects were enrolled in the study. However, only 189 subjects started and completed the study cute due to surgeries being cancelled, no Rocuronium given, missing data, or monitor malfunction.
Groups:
- Subjects Undergoing Elective Surgery Involving the Intraoperative Use of Rocuronium: Subjects undergoing elective surgery requiring neuromuscular blockade. Subjects all receive the neuromuscular blockade drug Rocuronium based on study protocol. Depending on depth of block (objectively assessed by TOF response), Neostigmine, Sugammadex, or no reversal drug is used to reverse block prior to extubation.
Period: Overall Study
Arm/Group | Subjects Undergoing Elective Surgery Involving the Intraoperative Use of Rocuronium
Started | 189
Completed | 189
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Subjects Undergoing Elective Surgery Involving the Intraoperative Use of Rocuronium
Number analyzed (Participants) | 189
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 162
  >=65 years | 27
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 71
  Male | 118
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 11
  Asian | 4
  Native Hawaiian or Other Pacific Islander | 3
  Black or African American | 19
  White | 152
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 189

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Postoperative Residual Neuromuscular Blockade at Time of Extubation
Description: Train-of-four ratio <0.9 as measured by electromyography or <1.0 measured by acceleromyography
Time Frame: Within two minutes of extubation
Measure: Count of Participants; unit: Participants
Arm/Group | Subjects Undergoing Elective Surgery Involving the Intraoperative Use of Rocuronium
Number analyzed (Participants) | 189
Participants | 0

2. Secondary Outcome: Incidence of Severe Postoperative Residual Neuromuscular Blockade at Time of Extubation
Description: Train-of-four ratio <0.7 as measured by electromyography
Time Frame: Within two minutes of extubation
Measure: Count of Participants; unit: Participants
Arm/Group | Subjects Undergoing Elective Surgery Involving the Intraoperative Use of Rocuronium
Number analyzed (Participants) | 189
Participants | 0

ADVERSE EVENTS:
Time Frame: Adverse event data was collected through the study duration which was for less than 1 day (from the beginning of surgery to discharge from the PACU after surgery).
Arm/Group | Subjects Undergoing Elective Surgery Involving the Intraoperative Use of Rocuronium
All-Cause Mortality (participants affected / at risk) | 0/189
Serious Adverse Events (participants affected / at risk) | 0/189
Other Adverse Events (participants affected / at risk) | 0/189

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2019-05-08): https://cdn.clinicaltrials.gov/large-docs/01/NCT03958201/Prot_001.pdf
  • Statistical Analysis Plan (2019-05-08): https://cdn.clinicaltrials.gov/large-docs/01/NCT03958201/SAP_002.pdf
  • Informed Consent Form (2019-05-08): https://cdn.clinicaltrials.gov/large-docs/01/NCT03958201/ICF_003.pdf